CLINICAL TRIAL: NCT05720494
Title: Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Doses of JZP441 in Healthy Adult Participants: A Double-Blind, Randomized, Placebo-Controlled Phase 1 Study
Brief Title: A Multiple Ascending Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics of JZP441 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JZP441-102
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Healthy Participants
Keywords: Healthy Participants; JZP441

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JZP441 (Experimental): Healthy participants who will be randomized to receive an oral dose of JZP441.
  Interventions: Drug: JZP441
- Placebo (Placebo Comparator): Healthy participants who will be randomized to receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JZP441 — Oral study drug administered for up to 4 weeks
  Arms: JZP441
Drug: Placebo — Oral placebo administered for up to 4 weeks
  Arms: Placebo

SUMMARY:
Treatments for narcolepsy and hypersomnolence disorders should have good oral bioavailability and brain penetration properties. JZP441 has demonstrated wake-promoting efficacy and anticataplectic activity in nonclinical studies and may represent a novel approach for these patients.

DETAILED DESCRIPTION:
This Phase 1, double-blind, randomized, placebo-controlled, parallel group study is designed to characterize the safety, tolerability, and PK of multiple ascending doses of JZP441 for up to 4 weeks in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Is 18 to 50 years of age inclusive, at the time of signing the informed consent
* Are overtly healthy as determined by medical evaluation, including medical history, physical exam, laboratory tests, and cardiac/blood pressure monitoring.

Exclusion Criteria:

* History or presence of gastrointestinal (including prior bariatric bypass surgery), hepatic or renal disease, or any other condition that, in the investigator opinion, may interfere with absorption, distribution, metabolism, or excretion of drugs
* Presence of renal impairment or calculated eGFR < 80 mL/min/1.73 m^2.
* Triplicate 12-lead ECG demonstrating a mean QTcF > 450 msec for males and > 470 msec for females or any other clinically significant ECG abnormality per investigator assessment prior to dose of study intervention
* Presence or history of significant cardiovascular disease including (but not limited to): myocardial infarction, uncontrolled hypertension, systolic BP ≥ 140 mmHg or diastolic BP ≥ 90 mmHg (at Screening or baseline consistent with protocol specifications), angina pectoris, clinically significant arrhythmias, clinically significant valvular heart disease, history of any revascularization procedures or second or third degree heart block with/without a pacemaker, heart failure, or family history of Torsades de Pointes
* Current diagnosis of or receiving treatment for depression; past (within 5 years) clinically significant major depressive episode; history of suicide attempt, current suicidal risk as determined from history, or presence of active suicidal ideation as indicated by a positive response to item 4 or item 5 on the C-SSRS (within the past 6 months)
* History or presence of bipolar disorder, bipolar related disorders, schizophrenia, schizophrenia spectrum disorders, or clinically significant psychiatric disorders, including other psychotic disorders
* History (within past 2 years at Screening) or presence of substance use disorder (including alcohol) or seeking treatment for alcohol or substance abuse related disorder
* History of seizure disorder or a physical condition that would increase seizure risk
* History of head trauma or concussions that are deemed clinically significant by the investigator
* Have used tobacco products or products for smoking cessation within 90 days before screening, including nicotine-containing products, or history of significant use of tobacco (> 10 cigarettes or equivalent per day) within 1 year before Screening, or unwilling to refrain from nicotine-containing products for the duration of the study
* Participants who are taking a concomitant medication or supplement that lowers seizure threshold (eg, kratom)
* Participants who have recently (< 2 weeks) discontinued a drug or supplement for which discontinuation would lower seizure threshold (eg, benzodiazepine medication)
* Participation in a previous JZP441 clinical study
* Positive alcohol test or urine drug screen (including cannabinoids and cotinine) at Screening or at any point throughout the duration of the study
* Presence at Screening of HIV antibody, Hepatitis B surface antigen, Hepatitis C antibody, or a clinical history of these infections
* History of clinically significant acute or chronic insomnia within the last 5 years

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Events | Day 1 up until 38 days after last dose of study drug, up to approximately 2 months
Pharmacokinetic Parameter Maximum Plasma Concentration (Cmax) Levels of JZP441 | Pre-dose and multiple post-dose timepoints, up to Day 28
Pharmacokinetic Parameter Time to Maximum Plasma Concentration (Tmax) of JZP441 | Pre-dose and multiple post-dose timepoints, up to Day 28
  Time to maximum plasma concentration (Tmax), time of maximum observed plasma concentration post first dose but before second dose during the 24-hour dosing interval (Tmax1), and time of maximum observed plasma concentration post second dose during the 24-hour dosing interval (Tmax2), and time of last quantifiable concentration (Tlast) will be assessed.
Pharmacokinetic Parameter Terminal Elimination Half-life (T1/2) of JZP441 | Pre-dose and multiple post-dose timepoints, up to Day 28
Pharmacokinetic Parameter Area Under the Concentration-Time Curve (AUC) of JZP441 | Pre-dose and multiple post-dose timepoints, up to Day 28
  Area under the concentration-time curve from time 0 to 24 hours (AUC0-24), area under the concentration-time curve from time zero to time of the last quantifiable concentration (AUC0-last), and area under the concentration-time curve from time zero extrapolated to infinity (AUC∞) will be assessed.
Pharmacokinetic Parameter Apparent Oral Clearance (CL/F) of JZP441 | Pre-dose and multiple post-dose timepoints, up to Day 28
Pharmacokinetic Parameter Apparent Volume of Distribution (Vz/F) of JZP441 | Pre-dose and multiple post-dose timepoints, up to Day 28
Pharmacokinetic Parameter Accumulation Ratio of JZP441 | Pre-dose and multiple post-dose timepoints, up to Day 28
  Accumulation ratio (Cmax) and accumulation ratio (AUC) will be assessed.
Dose Proportionality of JZP441 for Maximum Concentration (Cmax) | Pre-dose and multiple post-dose timepoints, up to Day 28
  Dose proportionality of maximum concentration (Cmax), maximum observed plasma concentration post first dose but before second dose during the 24-hour dosing interval (Cmax1), and maximum observed plasma concentration post second dose during the 24-hour dosing interval (Cmax2) will be assessed.
Dose Proportionality of JZP441 for Area Under the Concentration-Time Curve (AUC) | Pre-dose and multiple post-dose timepoints, up to Day 28
  Dose proportionality of area under the concentration-time curve from 0 to 24 hours (AUC[0-24]) will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site 1, Salt Lake City, Utah, United States